CLINICAL TRIAL: NCT05609539
Title: Clinical Effectiveness of an Off-the-shelf Single REnal Scalloped sTent-graft for HOstile NEck Infrarenal Abdominal Aortic Aneurysm: Clinical Pivotal Trial
Brief Title: Clinical Effectiveness of an Off-the-shelf Single REnal Scalloped sTent-graft for HOstile NEck Infrarenal Abdominal Aortic Aneurysm
Acronym: RESTHONE
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Collaborators: Ospedale di Circolo - Fondazione Macchi (Other); Azienda Ospedaliera di Padova (Other); Azienda Ospedaliera Ordine Mauriziano di Torino (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Roberto Silingardi, MD, Medical Doctor, Azienda Ospedaliero-Universitaria di Modena
Other Study IDs: RESTHONE
Record Dates: First submitted 2022-10-31; First posted 2022-11-08 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: AAA; EVAR; Hostile Neck Anatomy
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- AAA patients with a mismatched takeoff of the renal arteries candidated to standard EVAR: Patients suffering to AAA with a mismatched takeoff (>10mm) of the renal arteries
  Interventions: Device: Endovascular Aortic Repair (EVAR)

INTERVENTIONS:
Device: Endovascular Aortic Repair (EVAR) — Techniques for delivery and deployment of the standard device have been well described by different papers, but for the "prototype" some attention is required.
  Once the device was advanced at the level of the lowest RA the C-Arm has been moved to correct the parallax effect and positioned orthogonally to the origin of the artery. This procedure permits perfectly matching the scallop with the artery takeoff.
  A selective angiogram was performed to assure the patency of the lower RA. After the deployment of the main body proper iliac extensions were delivered to completely exclude the aneurysm as standard practice.

SUMMARY:
The goal of this multicenter, observational cohort study is to evaluates the clinical effectiveness of a single-renal scallop custom-made stent-graft (TREO, Terumo Aortic, Sunrise, FL) to treat "hostile" AAA with mismatched renal arteries as actual standard of care in this Vascular Unit The main question it aims to answer are: if a dedicated devices could improve the results in the endovascular treatment of patients suffering to infrarenal abdominal aortic aneurism with a mismatched takeoff of the renal arteries.

Participants responding to inclusion criteria will be treated as best clinical practice with a custom made device with a single scallop for the renal artery. The minimum follow-up requested, as standard clinical practice, was: 3-months, 12-18 months- and 5-years CTA; clinical and DUS examination at 6- and 12- and 36-months after the intervention and yearly thereafter.

No comparison group was present.

DETAILED DESCRIPTION:
Endovascular aneurysm repair (EVAR) is currently the preferred choice to treat the abdominal aortic aneurysms (AAA) with a feasible anatomy. However, approximately 40-60% of AAA patients presented unfavorable characteristics for EVAR, mainly due to a "hostile neck anatomy". In ''real-world'' clinical practice, up to 44% of EVAR cases are performed outside Instruction For Use (IFU) for an adverse neck anatomy6. Short (<15-mm), angulated (>60°), and wide (>28-mm) aortic necks are the main features concurring to the proximal HNA.

The recourse to standard EVAR is currently routine for patients who are not eligible for OR, with acceptable short- and mid-term outcomes, but the long-term durability of EVAR depends on maintaining proper sealing between the endograft and the aortic neck as well as the iliac arteries. HNAs demonstrated worse results when compared to "favorable" ones in terms of technical success (94% vs. 98%) and type-Ia endoleak rate (10% vs. 2%). The issue linked to an unfavorable anatomy can be addressed with more complex techniques, but these are limited by high production costs and considerable complexity .

TREO (Terumo Aortic, Inchinnan, Renfrewshire, UK; formerly Treovance, Bolton Medical, Sunrise, Fla) is a standard bifurcated, modular stent-graft that has shown compelling early- and mid-term results. It seems clear that several physicians are still looking for a feasible solution for HNA patients to keep the complexity of the procedure comparable to standard EVAR while yielding improved results.

Moreover, there is a lack of publications addressing the issue of mismatched take-off of the renal arteries (RAs). This morphology seems to influence the sealing length and could justify the introduction of dedicated devices. A recent study from our group currently under review for publication demonstrated that 25% of patients eligible for EVAR presented with mismatched RAs and that a dedicated device could improve sealing significantly. The study group sealing zone's length increased by about 25% when applying a hypothetical prototype with a single 10x10mm (wide x high) renal scallop. The same approach could be applied to the sealing surface with similar results. In the light of obtained results in selected patients, the use of a "single renal-scallop" custom-made device has been our standard of care.

The results will demonstrate whether the supra mentioned graft can the treatment of AAA with mismatched RAs in the real world. The effectiveness will be evaluated in terms of technical and clinical success.

The benefits could be relevant for the patients in terms of reduction of procedure-related adverse events such as endoleaks and related re-interventions. Furthermore, the use of custom-made standardized devices could significantly reduce costs for health care providers and in the future, it could be the base for an "off-the-shelf" endograft. Procedure-related complications were expected to be similar to standard EVAR and reduced in comparison with literature reporting adverse events in more complex techniques.

The present study aims to evaluate the clinical effectiveness of the custom-made standardized single renal scalloped stent-graft (Treo, Terumo Aortic) to treat infrarenal AAA. The final objective will be to employ the data obtained in this cohort for a future eventual development of an "off-the-shelf" device dedicated to patients with mismatched renal arteries. Such an endograft could keep the complexity of the procedure as similar as possible to standard EVAR while improving sealing.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by infrarenal AAA > 50mm
* Treated in election for non-symptomatic AAA
* Anatomy inside Treo (Terumo Aortic) instruction to use (IFU)
* Distance between renal arteries >10mm on aortic center-lumen-line
* Age > 18
* Patient fit to plead
* Both sex
* Written informed consent
* Treated in the coordinator center or in one of the study's participating centers
* Minimum follow-up requested: 3-months, 12-18 months and 5-years CTA; clinical and DUS examination at 6- and 12- and 36-months after the intervention and yearly thereafter

Exclusion Criteria:

* Patients with aortic pathologies different from AAA (aortic ulcers, dissection, pseudo-aneurysm etc)
* Treated in urgent/emergent setting for symptomatic or ruptured AAA
* AAA < 50mm
* Outside TREO (Terumo Aortic) IFU
* With an inter-renal distance measured of the center-lumen-line <10mm
* Age <18
* Unfit to plead
* Refused to sign the informed consent
* Treated outside the coordinator centers or in one of the study's participating center's
* Refusal to adhere to the requested follow-up

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients fit to plead and with a diagnosis of AAA > 50mm with a mismatched takeoff of tthe renal arteries. All the patients must be fit to ever with a standard endoggraft and must be able to carry out adhere the follow-up requested
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-09-28 (Actual); Study Completion 2025-09-28 (Actual)

PRIMARY OUTCOMES:
Evaluation of the clinical effectiveness of the endovascular exclusion of infrarenal Abdominal Aortic Aneurysm with a single renal scallop endograft | up to 24 hours
  Clinical effectiveness measured in terms of technical and clinical success. Technical success was defined as successful introduction and deployment of the device in the absence of surgical conversion or mortality, type I or III endoleaks, or graft limb obstruction. A technical success thus implies the following qualifying details: 1. Successful access to the arterial system using a remote site; 2. successful deployment of the endoluminal graft with secure proximal and distal fixation; 3. absence of either a type I or III endoleak; 4. patent endoluminal graft without significant twist, kinks, or obstruction by intraoperative measurements; 5 patency of both renal arteries and at least one hypogastric artery.

SECONDARY OUTCOMES:
Evaluation of the intra-operative and peri-operative (within 30 days) adverse events | up to 30 days
Collection of eventual adverse events related to the treatment procedure and eventual post-hoc analysis | "through study completion, an average of 2 years".
Evaluation of reintervention rate | "through study completion, an average of 2 years".
Evaluation time elapsed from procedure to re-intervention | "through study completion, an average of 2 years".
Evaluation of the association between baseline and anatomical features to adverse technical success, clinical success and reintervention rate | "through study completion, an average of 2 years".
Evaluation of the average procedural time | up to 24 hours
Evaluation of the average fluoroscopy time | up to 24 hours
Evaluation of the average contrast medium (CM) | up to 24 hours
Evaluation of the average dose absorption (DAP) mGy/m3 | up to 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Silingardi, Prof., Study Chair — AOU di Modena
Locations (1):
- AOU di Modena, Baggiovara, Modena, Italy

REFERENCES:
- [Background] Marone EM, Freyrie A, Ruotolo C, Michelagnoli S, Antonello M, Speziale F, Veroux P, Gargiulo M, Gaggiano A. Expert Opinion on Hostile Neck Definition in Endovascular Treatment of Abdominal Aortic Aneurysms (a Delphi Consensus). Ann Vasc Surg. 2020 Jan;62:173-182. doi: 10.1016/j.avsg.2019.05.049. Epub 2019 Aug 6. PMID 31394211
- [Background] Muhs BE, Jordan W, Ouriel K, Rajaee S, de Vries JP. Matched cohort comparison of endovascular abdominal aortic aneurysm repair with and without EndoAnchors. J Vasc Surg. 2018 Jun;67(6):1699-1707. doi: 10.1016/j.jvs.2017.10.059. Epub 2017 Dec 18. PMID 29248241
- [Background] Wanhainen A, Verzini F, Van Herzeele I, Allaire E, Bown M, Cohnert T, Dick F, van Herwaarden J, Karkos C, Koelemay M, Kolbel T, Loftus I, Mani K, Melissano G, Powell J, Szeberin Z, Esvs Guidelines Committee, de Borst GJ, Chakfe N, Debus S, Hinchliffe R, Kakkos S, Koncar I, Kolh P, Lindholt JS, de Vega M, Vermassen F, Document Reviewers, Bjorck M, Cheng S, Dalman R, Davidovic L, Donas K, Earnshaw J, Eckstein HH, Golledge J, Haulon S, Mastracci T, Naylor R, Ricco JB, Verhagen H. Editor's Choice - European Society for Vascular Surgery (ESVS) 2019 Clinical Practice Guidelines on the Management of Abdominal Aorto-iliac Artery Aneurysms. Eur J Vasc Endovasc Surg. 2019 Jan;57(1):8-93. doi: 10.1016/j.ejvs.2018.09.020. Epub 2018 Dec 5. No abstract available. PMID 30528142
- [Background] Chaikof EL, Dalman RL, Eskandari MK, Jackson BM, Lee WA, Mansour MA, Mastracci TM, Mell M, Murad MH, Nguyen LL, Oderich GS, Patel MS, Schermerhorn ML, Starnes BW. The Society for Vascular Surgery practice guidelines on the care of patients with an abdominal aortic aneurysm. J Vasc Surg. 2018 Jan;67(1):2-77.e2. doi: 10.1016/j.jvs.2017.10.044. PMID 29268916
- [Background] Speziale F, Sirignano P, Setacci F, Menna D, Capoccia L, Mansour W, Galzerano G, Setacci C. Immediate and two-year outcomes after EVAR in "on-label" and "off-label" neck anatomies using different commercially available devices. analysis of the experience of two Italian vascular centers. Ann Vasc Surg. 2014 Nov;28(8):1892-900. doi: 10.1016/j.avsg.2014.06.057. Epub 2014 Jul 7. PMID 25011083
- [Background] Stather PW, Wild JB, Sayers RD, Bown MJ, Choke E. Endovascular aortic aneurysm repair in patients with hostile neck anatomy. J Endovasc Ther. 2013 Oct;20(5):623-37. doi: 10.1583/13-4320MR.1. PMID 24093314
- [Background] AbuRahma AF, DerDerian T, AbuRahma ZT, Hass SM, Yacoub M, Dean LS, Abu-Halimah S, Mousa AY. Comparative study of clinical outcome of endovascular aortic aneurysms repair in large diameter aortic necks (>31 mm) versus smaller necks. J Vasc Surg. 2018 Nov;68(5):1345-1353.e1. doi: 10.1016/j.jvs.2018.02.037. Epub 2018 May 22. PMID 29802043
- [Background] Antoniou GA, Antoniou SA, Torella F. Editor's Choice - Endovascular vs. Open Repair for Abdominal Aortic Aneurysm: Systematic Review and Meta-analysis of Updated Peri-operative and Long Term Data of Randomised Controlled Trials. Eur J Vasc Endovasc Surg. 2020 Mar;59(3):385-397. doi: 10.1016/j.ejvs.2019.11.030. Epub 2019 Dec 30. PMID 31899100
- [Background] Sveinsson M, Sonesson B, Kristmundsson T, Dias N, Resch T. Long-term outcomes after fenestrated endovascular aortic repair for juxtarenal aortic aneurysms. J Vasc Surg. 2022 Apr;75(4):1164-1170. doi: 10.1016/j.jvs.2021.11.050. Epub 2021 Nov 25. PMID 34838610
- [Background] Eagleton MJ, Stoner M, Henretta J, Dryjski M, Panneton J, Tassiopoulos A, Mehta M, Pearce B, Sharafuddin MJ; TREO Investigators. Safety and effectiveness of the TREO stent graft for the endovascular treatment of abdominal aortic aneurysms. J Vasc Surg. 2021 Jul;74(1):114-123.e3. doi: 10.1016/j.jvs.2020.10.083. Epub 2020 Nov 28. PMID 33253871
- [Background] D'Oria M, Galeazzi E, Veraldi GF, Garriboli L, Sacca S, Farneti F, Mezzetto L, Mastrorilli D, Lepidi S; ITA-ENDOBOOT registry collaborators.. Impact of Proximal Neck Anatomy on Short-Term and Mid-Term Outcomes After Treatment of Abdominal Aortic Aneurysms With New-Generation Low-Profile Endografts. Results From the Multicentric "ITAlian North-East Registry of ENDOvascular Aortic Repair With the BOltOn Treo Endograft (ITA-ENDOBOOT)". Ann Vasc Surg. 2022 Mar;80:37-49. doi: 10.1016/j.avsg.2021.08.059. Epub 2021 Nov 6. PMID 34752851
- [Background] Murray D, Szeberin Z, Benevento D, Abdallah F, Palasciano G, Lescan M, Uberoi R, Setacci C. A comparison of clinical outcomes of abdominal aortic aneurysm patients with favorable and hostile neck angulation treated by endovascular repair with the Treovance stent graft. J Vasc Surg. 2020 Jun;71(6):1881-1889. doi: 10.1016/j.jvs.2019.07.096. Epub 2019 Nov 2. PMID 31690524
- [Background] Oderich GS, Farber MA, Schneider D, Makaroun M, Sanchez LA, Schanzer A, Beck AW, Starnes BW, Fillinger M, Tenorio ER, Chen M, Zhou Q; Zenith Fenestrated Study Investigators. Final 5-year results of the United States Zenith Fenestrated prospective multicenter study for juxtarenal abdominal aortic aneurysms. J Vasc Surg. 2021 Apr;73(4):1128-1138.e2. doi: 10.1016/j.jvs.2020.08.128. Epub 2020 Sep 3. PMID 32891806
- [Background] Gallitto E, Gargiulo M, Freyrie A, Mascoli C, Massoni Bianchini C, Ancetti S, Faggioli G, Stella A. The endovascular treatment of juxta-renal abdominal aortic aneurysm using fenestrated endograft: early and mid-term results. J Cardiovasc Surg (Torino). 2019 Apr;60(2):237-244. doi: 10.23736/S0021-9509.16.09049-2. Epub 2015 Sep 29. PMID 26417936
- [Background] Locham S, Faateh M, Dhaliwal J, Nejim B, Dakour-Aridi H, Malas MB. Outcomes and cost of fenestrated versus standard endovascular repair of intact abdominal aortic aneurysm in the United States. J Vasc Surg. 2019 Apr;69(4):1036-1044.e1. doi: 10.1016/j.jvs.2018.06.211. Epub 2018 Oct 3. PMID 30292604

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT05609539/Prot_SAP_000.pdf